CLINICAL TRIAL: NCT00987038
Title: A Phase 1, Open Label, Multiple Dose Study Of The Effect Of PF-04171327 On Midazolam Pharmacokinetics In Healthy Volunteers
Brief Title: A Midazolam Drug Interaction Study With PF-04171327
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9391007
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Healthy Volunteers
Keywords: drug interaction CYP3A4 glucocorticoids midazolam
MeSH Terms: interventions — fosdagrocorat; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04171327 and Midazolam (Other)
  Interventions: Drug: PF-04171327 25 mg; Drug: Midazolam 2 mg

INTERVENTIONS:
Drug: PF-04171327 25 mg — One 25 mg tablet administered once a day for 15 days
Drug: Midazolam 2 mg — Midazolam oral syrup 2mg dose administered once on Day 1 and once on Day 15

SUMMARY:
The purpose of this study is to investigate the effects of multiple doses of PF-04171327 on the blood levels (pharmacokinetics) of midazolam

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and/or females (non-childbearing potential) volunteers.
* Cortisol level within normal reference range of the laboratory.

Exclusion Criteria:

* History of intolerance or significant adverse effect with glucocorticoid (steroid) therapy.
* History or current positive results for HIV, Hepatitis B or C or active TB or currently undergoing treatment for TB.
* Known history of hypersensitivity, allergy severe drug reaction or unable to tolerate midazolam or other benzodiazepines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUCinf of midazolam | 17 days

SECONDARY OUTCOMES:
AUClast, Cmax, Tmax, t1/2 | 17 days
Vital Signs, Clinical Laboratory tests and Adverse Events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Ripp SL, Mukherjee A, Eng H, Stock T, Fleishaker D, Checchio T, Tammara B. In Vitro and In Vivo Investigation of Potential for Complex CYP3A Interaction for PF-00251802 (Dagrocorat), a Novel Dissociated Agonist of the Glucocorticoid Receptor. Clin Pharmacol Drug Dev. 2018 Mar;7(3):244-255. doi: 10.1002/cpdd.411. Epub 2017 Nov 7. PMID 29112329
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9391007&StudyName=A%20Midazolam%20Drug%20Interaction%20Study%20With%20PF-04171327